CLINICAL TRIAL: NCT02561338
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled, 12-week Phase II Study to Evaluate the Safety, Tolerability, Efficacy and Population PK of HMS5552 in Type 2 Diabetic Adult Subjects
Brief Title: A Multi-center 12-week Study of HMS5552 in T2DM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hua Medicine Limited (Industry)
Collaborators: Tigermed Consulting Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HMM0201
Record Dates: First submitted 2015-09-23; First posted 2015-09-28 (Estimated); Results first posted 2020-03-10 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-02

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: GKA,T2DM,HMS5552
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Dorzagliatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- HMS5552 dose 1 (Experimental): 75mgQD oral administration
  Interventions: Drug: HMS5552
- HMS5552 dose 2 (Experimental): 100mgQD oral administration
  Interventions: Drug: HMS5552
- HMS5552 dose 3 (Experimental): 50mgBID oral administration
  Interventions: Drug: HMS5552
- HMS5552 dose 4 (Experimental): 75mgBID oral administration
  Interventions: Drug: HMS5552
- Placebo (Placebo Comparator): Placebo, BID/QD oral administration
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: HMS5552 — 75mgQD
  Other Names: GKA
  Arms: HMS5552 dose 1
Drug: HMS5552 — 100mgQD
  Other Names: GKA
  Arms: HMS5552 dose 2
Drug: HMS5552 — 50mgBID
  Other Names: GKA
  Arms: HMS5552 dose 3
Drug: HMS5552 — 75mgBID
  Other Names: GKA
  Arms: HMS5552 dose 4
Other: Placebo — QD/BID
  Arms: Placebo

SUMMARY:
This study evaluates the safety, tolerability, efficacy and population PK of HMS5552 in type 2 diabetic adult subjects,there will be 5 groups ,4 groups will receive HMS5552,while 1 will receive placebo.

DETAILED DESCRIPTION:
Glucokinase (GK, also called hexokinase IV or D) can phosphosphorylate glucose to glucose-6-phosphate (G-6-P) in pancreatic β-cells and liver cells, which represents the first step of glucose metabolism. GK also acts as a glucose sensor and exerts a key role in maintaining glucose homeostasis. HMS5552 is a 4th-generation GK agonist or activator (GKA), which was originally licensed from Roche and subsequently developed by Hua Medicine. HMS5552 has been shown to activate GK in pancreatic beta cells, liver and intestinal epithelial cells. It regulates systemic blood glucose through a variety of mechanisms including directly enhancing insulin release (pancreas), inhibiting production of endogenous glucose (liver) and by indirectly promoting GLP-1 release (enteroendocrine L-cells).

ELIGIBILITY:
Inclusion Criteria:

1. Male & female, 40~75 years old
2. T2DM patients，anti-hyperglycemic drug-naïve and on diet & exercise for at least 3 months, or with glucose controlled by Metformin or α-glucosidase inhibitor alone
3. HbA1c 7.5~10.5% at screening and pre-randomization
4. Fasting plasma glucose (FPG)7.0~11.1 millimole/liter (mmol/L, local lab) at screening, and 7.0~13.3 millimole/liter (mmol/L, central lab) at pre-randomization
5. BMI: 19~30kg/m^2 & TG<5.5mmol/L

Exclusion Criteria:

1. T1D，secondary DM, pre-DM
2. kidney diseases or eGFR MDRD<60ml/min/1.73m^2
3. unstable CVDs
4. liver diseases
5. mental or CNS diseases

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Actual)
Dates: Start 2015-09; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dalong Zhu, MD，PhD, Principal Investigator — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Locations (1):
- Nanjing Drum Tower Hospital The Affiliated Hospital of Nanjing University Medical School, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhu D, Gan S, Liu Y, Ma J, Dong X, Song W, Zeng J, Wang G, Zhao W, Zhang Q, Li Y, Fang H, Lv X, Shi Y, Tian H, Ji L, Gao X, Zhang L, Bao Y, Lei M, Li L, Zeng L, Li X, Hou X, Zhao Y, Hu T, Ge X, Zhao G, Li Y, Zhang Y, Chen L. Dorzagliatin monotherapy in Chinese patients with type 2 diabetes: a dose-ranging, randomised, double-blind, placebo-controlled, phase 2 study. Lancet Diabetes Endocrinol. 2018 Aug;6(8):627-636. doi: 10.1016/S2213-8587(18)30105-0. Epub 2018 May 4. PMID 29735394

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo, BID/QD
Period: Overall Study
Arm/Group | HMS5552 Dose 1 | HMS5552 Dose 2 | HMS5552 Dose 3 | HMS5552 Dose 4 | Placebo
Started | 53 | 50 | 51 | 51 | 53
Completed | 45 | 44 | 42 | 46 | 51
Not Completed | 8 | 6 | 9 | 5 | 2

BASELINE CHARACTERISTICS:
Population: In the group HMS5552 dose3, a subject without follow-up data for HbA1c available was excluded. And in the group HMS5552 dose4, two subjects without follow-up data for HbA1c available were excluded. So the overall number of baseline participants is not consistent with numbers provided in any of the rows in the participant flow module.
Groups:
- Placebo: Placebo: BID/QD
- Total: Total of all reporting groups
Arm/Group | HMS5552 Dose 1 | HMS5552 Dose 2 | HMS5552 Dose 3 | HMS5552 Dose 4 | Placebo | Total
Number analyzed (Participants) | 53 | 50 | 50 | 49 | 53 | 255
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.58 (9.159) | 56.7 (7.670) | 54.92 (8.137) | 55.42 (7.659) | 54.73 (8.499) | 55.88 (8.271)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 22 | 16 | 18 | 22 | 104
  Male | 27 | 28 | 34 | 31 | 31 | 151
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 53 | 50 | 50 | 49 | 53 | 255
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 53 | 50 | 50 | 49 | 53 | 255
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  China | 53 | 50 | 50 | 49 | 53 | 255
HbA1c [Mean (Standard Deviation); unit: percentage of glycated hemoglobin] | 8.44 (0.803) | 8.27 (0.639) | 8.33 (0.653) | 8.46 (0.670) | 8.39 (0.780) | 8.38 (0.712)
FPG [Mean (Standard Deviation); unit: mmol/L] | 9.933 (2.3356) | 9.127 (1.4868) | 9.390 (1.5317) | 9.859 (1.9902) | 9.277 (1.7608) | 9.518 (1.8663)
2h PPG [Mean (Standard Deviation); unit: mmol/L] | 18.042 (3.3004) | 17.429 (3.2023) | 17.243 (3.0943) | 17.884 (3.1303) | 16.950 (3.7282) | 17.509 (3.3052)
Body Mass Index (BMI) units: kg/m^2 [Mean (Standard Deviation); unit: kg/m^2] | 24.718 (2.8672) | 25.010 (2.9374) | 24.686 (2.3112) | 25.321 (2.5419) | 25.188 (2.6113) | 25.321 (2.5419)
Diagnosis time [Mean (Standard Deviation); unit: years] | 3.37 (4.053) | 3.24 (4.304) | 3.27 (4.220) | 2.82 (3.230) | 3.41 (4.195) | 3.23 (3.984)

OUTCOME MEASURES:

1. Primary Outcome: After 12-week Treatment, the Change From Baseline in HbA1c
Description: Assess the percentage of Hemoglobin A1c (HbA1c) changes at week 12. In the group HMS5552 dose3, a subject without follow-up data for HbA1c available was excluded. And in the group HMS5552 dose4, two subjects without follow-up data for HbA1c available were excluded. So the overall number of baseline participants is not consistent with numbers provided in any of the rows in the participant flow module.
Time Frame: Baseline and 12 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of glycated hemoglobin
Groups:
- HMS5552 Dose 2: HMS5552:100mgQD
- Placebo: Placebo:BID/QD
Arm/Group | HMS5552 Dose 1 | HMS5552 Dose 2 | HMS5552 Dose 3 | HMS5552 Dose 4 | Placebo
Number analyzed (Participants) | 53 | 50 | 50 | 49 | 53
Percentage of glycated hemoglobin | -0.39 [-0.64 to -0.16] | -0.65 [-0.92 to -0.38] | -0.79 [-1.06 to -0.52] | -1.12 [-1.39 to -0.86] | -0.35 [-0.60 to -0.10]

2. Secondary Outcome: Change From Baseline in 2hPPG
Description: Using a standard meal tolerance test, to assess 2-h postprandial glucose (2hPPG). In this test, subjects were received meals standardised by China National Cereals, which supplied by Oils and Foodstuffs Corporation and contained 353 kcal, 75 g carbohydrate, 1.48 g fat, and 8.0 g protein. Collect the blood samples to detect blood glucose 2 hours after starting the meal.
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | HMS5552 Dose 1 | HMS5552 Dose 2 | HMS5552 Dose 3 | HMS5552 Dose 4 | Placebo
Number analyzed (Participants) | 53 | 50 | 50 | 49 | 53
mmol/L | -4.669 (2.325) | -4.945 (3.387) | -3.898 (3.535) | -4.899 (3.921) | -1.987 (3.312)

3. Secondary Outcome: Change From Baseline in FPG
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | HMS5552 Dose 1 | HMS5552 Dose 2 | HMS5552 Dose 3 | HMS5552 Dose 4 | Placebo
Number analyzed (Participants) | 53 | 50 | 50 | 49 | 53
mmol/L | -0.307 (2.000) | -0.382 (1.602) | -0.758 (2.150) | -1.319 (2.258) | -0.801 (1.752)

4. Post Hoc Outcome: Change From Baseline in MMTT (Mixed Meal Tolerance Test) β-cell Function Index
Description: Disposition index, i.e DI, by the insulin secretion sensitivity index-2 (ISSI-2). This is an calculated value which represents the ability of a person's pancreatic beta cells to lower blood glucose. A higher number means the pancreas is better able to secrete insulin and improve glucose levels. HOMA IR is an index used to evaluate the individual's insulin resistance level. The HOMA-IR index of normal individuals is 1. With the increase of insulin resistance, HOMA-IR index will be higher than 1.
Time Frame: Baseline and week 12
Population: Both of disposition index and HOMA-IR could reflect the function of β cell.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | HMS5552 Dose 1 | HMS5552 Dose 2 | HMS5552 Dose 3 | HMS5552 Dose 4 | Placebo
Number analyzed (Participants) | 53 | 50 | 50 | 49 | 53
units on a scale
  Disposition Index: number analyzed (Participants) | 40 | 45 | 42 | 44 | 49
  Disposition Index | 0.292 [0.065 to 0.838] | 0.198 [-0.075 to 0.532] | 0.216 [0.008 to 0.532] | 0.140 [-0.010 to 0.580] | 0.080 [-0.061 to 0.265]
  HOMA-IR: number analyzed (Participants) | 41 | 45 | 43 | 44 | 49
  HOMA-IR | -0.530 [-1.770 to 0.260] | -0.520 [-2.050 to 0.150] | -0.550 [-1.930 to 0.260] | -1.185 [-2.485 to -0.385] | -0.680 [-1.650 to 0.280]

ADVERSE EVENTS:
Time Frame: From randomization to 7 days after 12-week treatment
Description: Note: Hypoglycemia in this study was collected and analyzed as Special attention event separated from the analysis of Any other Advance Event. The Number Affected by Hypoglycemia was not included in the Total Number Affected by Any Other (Not including Serious) Adverse Event Above the Frequency Threshold in the third table.
Arm/Group | HMS5552 Dose 1 | HMS5552 Dose 2 | HMS5552 Dose 3 | HMS5552 Dose 4 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/50 | 0/51 | 0/51 | 0/53
Serious Adverse Events (participants affected / at risk) | 1/53 | 1/50 | 1/51 | 0/51 | 0/53
Other Adverse Events (participants affected / at risk) | 16/53 | 21/50 | 13/51 | 18/51 | 15/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HMS5552 Dose 1 (N=53) | HMS5552 Dose 2 (N=50) | HMS5552 Dose 3 (N=51) | HMS5552 Dose 4 (N=51) | Placebo (N=53)
Right Achilles Tendon Rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lacunar Infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Right Cerebral Infarction Of Basal Ganglia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HMS5552 Dose 1 (N=53) | HMS5552 Dose 2 (N=50) | HMS5552 Dose 3 (N=51) | HMS5552 Dose 4 (N=51) | Placebo (N=53)
Upper Respiratory Tract Infection (Infections and infestations) | 6 (6) | 6 (6) | 1 (1) | 4 (5) | 3 (3)
Hyperuricaemia (Metabolism and nutrition disorders) | 3 (3) | 6 (6) | 3 (3) | 4 (4) | 2 (2)
Dizziness (Nervous system disorders) | 2 (4) | 4 (9) | 4 (6) | 0 (0) | 0 (0)
Protein Urine Present (Investigations) | 3 (3) | 2 (2) | 0 (0) | 2 (2) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 3 (3)
Blood Creatine Phosphokinase Increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 5 (5)
White Blood Cells Urine Positive (Investigations) | 1 (1) | 0 (0) | 2 (2) | 3 (3) | 1 (1)
Hepatic Function Abnormal (Hepatobiliary disorders) | 2 (2) | 1 (1) | 3 (3) | 0 (0) | 1 (1)
High Density Lipoprotein Decreased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 4 (4) | 1 (1)
Ventricular Extrasystoles (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (2) | 3 (3) | 0 (0) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 3 (8) | 2 (2) | 3 (3) | 3 (10) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes